CLINICAL TRIAL: NCT00182637
Title: A Phase II Study of Bortezomib (VELCADE®) in Patients With Relapsed or Refractory Cutaneous T-Cell Lymphoma (CTCL)
Brief Title: Bortezomib in Treating Patients With Relapsed or Refractory Cutaneous T-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000439458; UCLA-0405014-02; MILLENNIUM-VEL-04-103
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2016-01

CONDITIONS: Lymphoma
Keywords: recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bortezomib (Experimental)
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well bortezomib works in treating patients with relapsed or refractory cutaneous T-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rates (complete response and partial response) and duration of response in patients with relapsed or refractory cutaneous T-cell lymphoma treated with bortezomib.
* Determine the safety and tolerability of this drug in these patients.

OUTLINE: This is an open-label study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 1 month and then at least every 3 months for 2 years or until disease progression.

PROJECTED ACCRUAL: A total of 15-25 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cutaneous T-cell lymphoma, including mycosis fungoides/Sézary syndrome
* Stage IB-IV disease
* Relapsed or refractory disease OR intolerant to ≥ 1 prior systemic therapy
* Measurable disease by radiological imaging or clinical finding
* Age Over 18
* Performance status Karnofsky 70-100%
* Hematopoietic

  * WBC > 2,000/mm^3
  * Absolute neutrophil count > 1,500/mm^3
  * Platelet count > 75,000/mm^3
  * Hemoglobin > 8.0 g/dL
* Hepatic

  * Bilirubin < 2 times upper limit of normal (ULN)
  * AST and ALT < 3 times ULN
* Renal

  * Creatinine < 1.5 times ULN
  * Creatinine clearance ≥ 30 mL/min
* Negative pregnancy test
* Fertile patients must use effective contraception
* More than 3 months since prior high-dose chemotherapy
* More than 30 days since prior and no other concurrent investigational drugs

Exclusion Criteria:

* history of myelodysplastic syndromes
* evidence of CNS disease
* pregnant or nursing
* peripheral neuropathy ≥ grade 2
* hypersensitivity to bortezomib, boron, or mannitol
* serious medical condition or psychiatric illness that would preclude study participation
* concurrent immunotherapy
* concurrent chemotherapy
* concurrent steroid dose > 10 mg/day of prednisone or its equivalent
* concurrent radiotherapy
* concurrent surgery for the malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2004-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren C. Pinter-Brown, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib: administration of bortezomib
Period: Overall Study
Arm/Group | Bortezomib
Started | 5 (active/on treatment date)
Completed | 2 (off study date)
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate After 2 Courses of Treatment
Time Frame: 2 months
Population: Only two subjects completed the trial. Study closed early due to lack of enrollment. No analysis performed.
Groups:
- Bortezomib: bortezomib
Arm/Group | Bortezomib
Number analyzed (Participants) | 0

2. Secondary Outcome: Time to Progression
Time Frame: 2 years
Population: Only two subjects completed the trial. Study closed early due to lack of enrollment. No analysis performed.
Arm/Group | Bortezomib
Number analyzed (Participants) | 0

3. Secondary Outcome: Toxicity
Time Frame: 2 years
Population: Only two subjects completed the trial. Study closed early due to lack of enrollment. No analysis performed.
Arm/Group | Bortezomib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the time that subjects signed consent until 30 days post treatment. Time frame varied depending on the time that the subject was on study. Approximately 6-7 months.
Arm/Group | Bortezomib
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib (N=5)
Fatigue (General disorders) | 2 (2)
Decrease Appetite (General disorders) | 1 (1)
Hot Flushes (General disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insominia (General disorders) | 1 (1)
Pain extremities, chest (Cardiac disorders) | 1 (1)
neuropathy extremities (General disorders) | 2 (3)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
chills / cough cold symptoms (Infections and infestations) | 1 (1)
generalized itching (General disorders) | 1 (2)
Body Aches / Flu Symptoms (Infections and infestations) | 1 (1)
Sensitive Skin (General disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No